CLINICAL TRIAL: NCT03961854
Title: Evaluation of the Safety, Tolerability and Immunological Response to Lactobacillus Johnsonii N6.2 in Children and Adolescents With T1D
Brief Title: Lactobacillus Johnsonii in Children and Adolescents With T1D
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB201901369; 2-SRA-2019-811-M-B (Other Grant/Funding Number: Juvenile Diabetes Research Foundation); OCR22462 (Other: UF OnCore)
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: probiotics; genetics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, placebo-controlled clinical trial will be carried out with children and adolescents (8-less than 18 years old) with T1D
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Active Comparator): The probiotic group will receive a daily capsule with Lactobacillus johnsonii N6.2 1x109 CFUs. Participants will consume one capsule (treatment or placebo) daily for 24 weeks.
  Interventions: Drug: L. johnsonii Probiotic
- Placebo Group (Placebo Comparator): The placebo group will receive a capsule daily with dried skim milk (vehicle of the probiotic). Participants will consume one capsule (treatment or placebo) daily for 24 weeks.
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: L. johnsonii Probiotic — Participants will consume one capsule of L. johnsonii probiotic daily for 24 weeks.
  Arms: Probiotic Group
Drug: Placebo Capsule — Participants will consume one capsule of placebo capsule of dried skim milk daily for 24 weeks.
  Arms: Placebo Group

SUMMARY:
While genetics demonstrated a major risk factor for the development of type 1 diabetes (T1D), microbiota dysbiosis has been suggested as an elicitor in immunological tolerance and of beta cell autoimmunity. The probiotic Lactobacillus johnsonii N6.2 may prevent or restore the gut flora and show systemic impacts and adaptive immunity in the T1D population thereby preserving beta cell function.

ELIGIBILITY:
Inclusion Criteria:

* have confirmed T1D by physician diagnosis
* have normal values at screening for complete blood count (CBC) and complete metabolic profiles (with the exception of fasting glucose and HbA1c)
* are able to swallow a capsule
* are willing to complete weekly online questionnaires
* are willing to consume a probiotic
* are willing to provide stool samples throughout the study
* are willing to provide blood samples throughout the study
* are willing to take three stimulated C-peptide tests
* are able to access a computer with Internet throughout the study

Exclusion Criteria:

* being treated for any diseases or illnesses such as gastrointestinal disease (gastric ulcers, Crohn's disease, ulcerative colitis, etc.)
* being treated for chronic kidney disease
* have had or are currently being treated for other immune-compromising diseases or conditions (HIV, AIDS, hepatitis, cancer, leukemia, organ transplant, Lupus, DiGeorge syndrome, selective deficiency of IgA, Bruton's disease etc.)
* have an underlying structural heart disease
* currently live with an immunocompromised person
* are currently taking medications for constipation and/or diarrhea
* have taken antibiotics within the past 2 weeks prior to randomization
* are currently taking a probiotic supplement and are unwilling to discontinue it a minimum of 2 weeks prior to the study start
* are a current smoker
* are currently pregnant or lactating or a female who plans to become pregnant in the next 6 months
* have a known allergy to milk or milk protein.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Safety will be evaluated according to complete blood count (CBC) and complete comprehensive metabolic panel (CMP) | 52 weeks
  CBC and CMP will be evaluated at four different time points during study: 1st measure will be at screening visit and before starting intervention (visit 1/week -4, baseline period), 2nd measure will be after 12 weeks after starting intervention (visit 2/ week 12), 3rd measure will be after the 24 weeks of intervention (visit 3/ week 24) and the 4th measure will be 24 weeks later, end of washout period (visit 4/week 48). Values should be within the normal values except for glucose.
Tolerance will be evaluated according to their responses on weekly questionnaires | 52 weeks
  The weekly questionnaire will ask participants to respond to questions regarding their gastrointestinal health (bowel movement frequency, gastrointestinal and other symptoms (i.e., constipation, diarrhea, stomach pain) and general wellness (if you consumed an antibiotic, visited a doctor, etc.). The questionnaires follow a scale from 1-7, 1 = No discomfort at all, 7 = Very severe discomfort.
Adverse Event and/or Serious Adverse Event | 24 weeks
  Adverse Event and/or Serious Adverse Event will be recorded daily by parents and notified to investigator within 24 hrs., in particular gastro-intestinal symptoms, fever and rashes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haller, Principal Investigator — University of Florida
Locations (1):
- UF Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No